CLINICAL TRIAL: NCT01501942
Title: A Double-blind, Placebo-controlled, Cross-over Study to Evaluate the Efficacy, Safety, Tolerability, Pharmacodynamics and Pharmacokinetics of Oral Administration of AIM-102 in Patients With Mild to Moderate Allergic Asthma
Brief Title: Efficacy, Safety, Tolerability, Pharmacodynamics and Pharmacokinetics of Oral Administration of AIM-102 in Patients With Mild to Moderate Allergic Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AIM Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: AIM102-201
Record Dates: First submitted 2011-12-26; First posted 2011-12-30 (Estimated); Last update posted 2014-02-14 (Estimated); Status verified 2014-02

CONDITIONS: Asthma
Keywords: Asthma; Allergen induced asthma; ATS Criteria (1)
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental): The active drug product is an oral solution of AIM-102 in phosphate buffered saline at a concentration of 35.0 mg/ml.
  Interventions: Drug: AIM-102, D-cyclohexylalanine-D-glutamic-glycine tripeptide
- Inactive product (Placebo Comparator): The matching placebo is an oral solution of phosphate buffered saline
  Interventions: Drug: Buffered Saline

INTERVENTIONS:
Drug: AIM-102, D-cyclohexylalanine-D-glutamic-glycine tripeptide — AIM-102 is supplied as an oral solution. Dose is 15 mg of AIM-102 per kg of patient weight measured on Treatment Day 1 of each treatment phase The study drug will be administered for 4 consecutive days with at least a 2 week wash-out period prior to crossing over to the alternative treatment for 4 days.
  Arms: Active
Drug: Buffered Saline — The matching placebo is an oral solution of phosphate buffered saline
  Arms: Inactive product

SUMMARY:
This is a Phase II, double-blind, placebo-controlled, cross-over trial to evaluate the efficacy of AIM-102 for the treatment of allergen-induced asthma. Individuals with stable, mild to moderate allergic asthma by American Thoracic Society (ATS) criteria (1), with a history of episodic wheeze and shortness of breath, will be eligible for enrollment.

The patients will receive 4 consecutive days of dosing of AIM-102 or placebo (inactive product) with an allergen challenge on day 3 of dosing to see how the patient's lung function is changed by using AIM-102 or placebo.

DETAILED DESCRIPTION:
This is a Phase II, double-blind, placebo-controlled, cross-over trial to evaluate the efficacy of AIM-102 for the treatment of allergen-induced asthma. Individuals with stable, mild to moderate allergic asthma by American Thoracic Society (ATS) criteria (1), with a history of episodic wheeze and shortness of breath, will be eligible for enrollment.

The study is divided into 2 parts.

Part 1: Screening

Patients who meet all entry criteria will be screened with a history, physical examination, spirometry, and routine laboratory tests. If they continue to meet entry criteria, their atopic status will be documented by skin testing against common airborne allergens (including cat, dust mite, grass, pollen). Twenty-four (24) hr later, an allergen challenge will be performed to confirm the presence of an Early Asthmatic Response (EAR) and Late Asthmatic Response (LAR). Methacholine PC20 and sputum differentials will be performed before and after allergen challenges. Only patients with a documented early and late asthmatic response to inhaled incremental allergen challenge will be eligible for entry into Part 2 of the study.

Part 2: Dosing and Follow-up

Patients will be assigned to receive drug and placebo in a random order, with at least a two week washout between treatment periods. Spirometry, vital signs, and asthma symptomatology, methacholine challenge, sputum differentials will be evaluated before the first dose and again 24 hr before allergen challenge. Allergen challenge will be performed in the morning of Day 3 of dosing, post-dose, with spirometry measured until seven hr post-challenge. Sputum will also be induced at seven hr following the allergen challenge. Methacholine challenge and sputum induction will be performed 24 hr after allergen challenges. Any adverse events (AEs) and asthma symptoms will be evaluated at each clinic visit. A physical examination, vital signs, ECG, spirometry and laboratory tests will be repeated at the termination visit.

ELIGIBILITY:
Inclusion Criteria:

The following inclusion must be met for study entry (Part 1 - Screening):

* Males and females between ≥ 18 and ≤ 65 years of age.
* Able and willing to provide written informed consent to participate in the study, in accordance with ICH GCP requirements.
* Non or ex-smoker, defined by an ex-smoker is defined as someone who completely stopped smoking for at least 12 months before Visit 1 of this study.
* Able to adhere to study procedures.
* In good general health without clinically significant medical history (see also Exclusion criteria below).
* Physical examination and laboratory results within the normal ranges, if not within the ranges, they must be without clinically significance within 28 days prior to dosing.
* Available for follow-up for the duration of the study (i.e. up to 10 weeks, including the Screening and Treatment Phases).
* Mild to moderate, stable, allergic asthma by the ATS criteria (1)
* History of episodic wheeze and shortness of breath; FEV1 at baseline at least 70% of the predicted value
* Males agree to practice adequate contraception throughout the duration of the study and up to one month after drug administration.

FEMALE-SPECIFIC INCLUSION CRITERIA:

* All females must have a negative serum pregnancy test at Screening Days -5 to -1 (Visit 5) and a negative urine pregnancy test at Day 1 of each Treatment Phase prior to dosing (Visits 6 and 11).
* A female patient must meet one of the following criteria:

  * No reproductive potential, defined as: menopausal for at least two years or surgically sterile for at least six months (i.e. has undergone hysterectomy, bilateral oophorectomy or tubal ligation) OR
  * Participant agrees to be heterosexually inactive from Screening Visit 1 until one month post final dose OR
  * Participant agrees to consistently practice adequate contraception from Screening Visit 1 until one month post final dose by one of the following methods, two methods must be used if hormonal contraception is used: Contraceptive pills (stable dose for at least 2 months prior to dosing on Day 1 (Visit 6) or patch, Norplant or Provera; intrauterine device (IUD), condom with spermicide or diaphragm (cervical cap) with spermicide.

In addition the inclusion criteria above, the following inclusion criteria must be met for entry into the Dosing Phase (Part 2):

* Positive methacholine challenge (PC20 ≤ 16 mg/ml)
* Positive skin-prick test to common aeroallergens (including cat, dust mite, grass, pollen)
* Positive allergen-induced early and late airway bronchoconstriction

Exclusion Criteria:

A patient will be excluded if one or more of the following conditions apply.

FEMALE ONLY EXCLUSIONS:

* Females who are pregnant or are lactating
* Females of childbearing potential who refuse to use an acceptable contraceptive regimen throughout the entire duration of the study (from the Screening visit until study completion) and for one month post dosing

RELEVANT MEDICAL HISTORY:

* Use of any nicotine containing products within 12 months prior to Screening or a smoking history > 10 pack years
* A worsening of asthma or a respiratory tract infection within 6 weeks preceding study entry
* Clinically significant and relevant abnormal findings in the clinical history, physical examination, ECG, or laboratory tests during Screening that would interfere with the objectives of the study or that would in the Investigator's opinion preclude safe completion of the study. Abnormal clinical history and/or findings could include:

  * Presence of significant gastrointestinal, liver or kidney disease, or any other conditions known to interfere with the absorption, distribution, metabolism or excretion of drugs or known to potentiate or predispose to undesired effects
  * Presence of significant cardiovascular, pulmonary, hematologic, neurological, psychiatric, endocrine, immunologic or dermatologic disease
  * Presence of out-of-range cardiac interval (PR < 110 msec, PR > 200 msec, QRS < 60 msec, QRS > 110 msec and QTc > 440 msec) on the screening ECG or other clinically significant ECG abnormalities
  * Autoimmune disease or immunodeficiency
  * History of clinically significant hypotensive episodes or symptoms of fainting, dizziness, or lightheadedness
  * Abnormal chest X-ray either at or within 1 year of Screening
  * Current acute or chronic illness (including infection) or recent recovery from acute illness which could, in the opinion of the Investigator, alter immune cell function (e.g., flu, cold or other respiratory infection, etc.)
  * Presence of a transplanted tissue or organ
  * Any evidence of malignancy [active and/or treated] within the previous five years or malignancy that is likely to recur during the period of the study
  * History of diabetes mellitus (Type I or II)
  * Thyroid disease (including thyroidectomy), requiring medication within the past 12 months
  * Asthma that is unstable or required emergent/urgent care, hospitalization or intubation during the past two years or that requires the use of oral or intravenous corticosteroids
  * Bleeding disorders (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions)
  * Major surgical procedure or significant traumatic injury within 12 months prior to the study treatment administration, OR minor surgery within one month prior to the study treatment administration or anticipation of the need for any surgery during the course of the study
  * Any other significant concomitant illness or injury that would interfere with the patient's participation in the study
  * Any clinically significant illness in the previous 28 days before the first day of dosing in either of the Treatment Phases of this study
  * Use of any enzyme-modifying drugs, including strong inhibitors of cytochrome P450 (CYP) enzymes (such as cimetidine, fluoxetine, quinidine, erythromycin, ciprofloxacin, fluconazole, ketoconazole, diltiazem and HIV antivirals) and strong inducers of CYP enzymes (such as barbiturates, carbamazepine, glucocorticoids, phenytoin, rifampin and St John's Wort), in the previous 30 days before Day 1 of this study
  * History of drug abuse including marijuana, PCP, cocaine, crack, LSD or other identified street drugs
  * Positive results to HIV, HbsAg or anti-HCV tests at Screening
  * Lung disease other than mild to moderate allergic asthma
  * Concomitant disease or condition which could interfere with the conduct of the study, or for which the treatment might interfere with the conduct of the study, or which would, in the opinion of the Investigator, pose an unacceptable risk to the patient in this study, including, but not limited to, cancer, alcoholism, drug dependency or abuse, or psychiatric disease
  * Recent (less than 1 year) history of alcohol dependency
* Any other medical, social, or geographical factor, which would make it unlikely that the patient will comply with study procedures (e.g. history of non-compliance)

PROHIBITED MEDICATION USE

* Systemic immunosuppressive or cytotoxic drug therapy (systemic corticosteroids, cyclophosphamide, methotrexate, cyclosporine, azathioprine, etc.) taken within two months prior to the study treatment administration. Corticosteroid nasal spray (e.g. for allergic rhinitis) or inhaled corticosteroid must have a 30 day washout prior to randomization (Visit 6)
* Significant history of drug dependency or alcohol abuse (> 3 units of alcohol per day, intake of excessive alcohol, acute or chronic)
* Use of any investigational therapy or participation in another clinical study within 30 days prior to the study drug administration
* Use of nonsteroidal anti-inflammatory drugs (NSAIDs) within 48 hr of dosing or aspirin within seven days of dosing and any time during the Treatment Phases
* Have chronic use of any other medication for treatment of allergic lung disease other than short-acting ß2-agonists or ipratropium bromide
* Use of caffeine-containing products or medications for 12 hr or alcohol or over the counter drugs including cold and allergy medications for 48 hr or inhaled bronchodilators for 8 hr prior to methacholine and allergen challenges

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2012-02; Primary Completion 2013-02 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline of the allergen-induced late asthmatic response (LAR) between AIM-102 and placebo. | Pre dose(s) and post dose(s) and 7 and 24 hours post allergen challenge
  Spirometry and the presence and severity of asthma symptoms will be assessed immediately before and immediately after each dose. Baseline and allergen-induced methacholine PC20, allergen-induced bronchoconstriction and allergen-induced airway inflammation will be assessed.
  AUC and maximum decrease in FEV1 for the late response will be compared between treatments using a one-way analysis of variance for the effects of treatment.

SECONDARY OUTCOMES:
Early Asthmatic Response | Pre-dose(s) and post-dose(s) and 3 hours after allergen challenge
  Spirometry & the presence and severity of asthma symptoms will be assessed immediately before and immediately after each dose. Baseline and allergen-induced methacholine PC20, allergen-induced bronchoconstriction and allergen-induced airway inflammation will be assessed.
  Allergen-induced increase in airway responsiveness is assessed by measuring the log methacholine PC20 difference from 24 hours before to 24 hours after allergen challenge.
• Comparison of the allergen-induced changes in sputum eosinophils at 7 hr and 24 hr post allergen, between the AIM-102 and placebo | Pre-dose and post-dose(s) and 7 and 24 hours post allergen challenge
  Allergen-induced sputum eosinophils will be compared between treatments using a two-way analysis of variance for the effects of treatment and time.
Comparison of allergen-induced inflammatory mediators at 7 hr and 24 hr post allergen, between AIM-102 and placebo. | Pre-dose and post-dose(s) and 7 and 24 hours post allergen challenge
  The allergen-induced airway inflammatory cells will be compared between treatments using a two-way analysis of variance.
Comparison of the allergen-induced airway hyperresponsiveness at 24 hours (hr) post allergen, between AIM-102 and placebo | Pre-dose and 24 hours post allergen challenge
  The allergen-induced airway hyperresponsiveness will be compared between treatments using a one-way analysis of variance for the effects of treatment.
To determine the pharmacokinetic (PK) profile of AIM-102 in normal healthy mild to moderate asthmatic patients upon repeat dosing of AIM-102 | Pre-dose for dosing Days 1, 2, 3, 4, & an optional Day 5, additional samples on Day 3 post-dose & allergen challenge,pre-dose, 1.5, 3, 4.5, 6, & 7.5 hr post-dose
  Drug plasma concentration data will be analyzed using a non-compartmental approach to obtain the following PK parameters:
  * peak plasma concentration
  * time to peak plasma concentration
  * elimination rate constant
  * terminal or elimination half-life
  * area under the concentration time curve from time 0 to last quantifiable concentration
  * area under the concentration time curve from time 0, extrapolated to infinity
  * oral clearance
  * oral volume of distribution

CONTACTS AND LOCATIONS:
Overall Officials: Paul O'Byrne, MD, Principal Investigator — McMaster University
Locations (2):
- Canada (2):
  - McMaster University, Hamilton, Ontario
  - Institut de cardiologie et de pneumologie de l'Hôpital Laval, Laval, Quebec